CLINICAL TRIAL: NCT06828133
Title: Egyptian Physical Therapists' Perceptions of Tele- Rehabilitation: an Online Open Survey on Acceptability, Preferences, and Needs
Brief Title: Egyptian Physical Therapists' Perceptions of Tele- Rehabilitation
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtihal Abdelaal Eissa Ali, researcher physiotherapist, Cairo University
Other Study IDs: P.T.REC/012/005612
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Acceptability, Preferences, and Needs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- observithional study of this group: observitional of this study

SUMMARY:
The healthcare industry has undergone a significant transformation with the integration of digital technologies, and one of the notable advancements in this field is tele-rehabilitation. Tele-rehabilitation, a subset of telehealth, involves the use of digital platforms to deliver physical therapy services remotely. This innovative approach allows healthcare providers to extend their reach, offering therapy to patients who might otherwise face barriers to accessing care,tele-rehabilitation has been recognized for its numerous benefits. It enhances access to physical therapy services, particularly for individuals living in remote or underserved areas. By reducing the need for travel, tele-rehabilitation offers significant convenience to patients, enabling them to receive therapy in the comfort of their homes.

ELIGIBILITY:
* Must be a licensed physical therapist with at least 3 years of experience practicing in Egypt.
* Must be 25 years of age or older.
* Must have access to the internet and be able to complete an online survey.
* Available to complete all survey-related questions.

Exclusion Criteria:

* Not currently practicing as a physical therapist.
* Diagnosed with conditions that impair the ability to complete an online survey.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: both male and female age between equale and more 25
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
acceptability | 6 months
  questionnaire

SECONDARY OUTCOMES:
preferences | 6 month
  quthionnaire

OTHER OUTCOMES:
needs | 6 mnoth
  quthionnaire

IPD SHARING:
Plan to Share IPD: Undecided